CLINICAL TRIAL: NCT05336227
Title: A Pilot Trial of Telehealth Active Video Gaming Using Immersive Virtual Reality on Cardiometabolic Health Among Youth With Cerebral Palsy
Brief Title: Telehealth Virtual Reality Gaming on Cardiometabolic Health Among Youth With Cerebral Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Byron Lai, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 300007833; 1R03HD107598-01 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
Keywords: physical activity; exercise; telehealth
MeSH Terms: conditions — Cerebral Palsy; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: One group that immediately receives the intervention. Another group that waits before receiving the same intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blinded to group allocation (data entry and analysis personnel).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Start - Virtual Reality Exergaming (Experimental): 12 weeks of virtual reality active video gaming using immersive commercially available equipment, with adapted games for people to play in the seated position. Maintain normal eating/nutritional behaviors.
  Interventions: Behavioral: Virtual Reality Exergaming
- Wait-list Control (No Intervention): Maintain habitual physical activity levels for 12 weeks, before receiving the same intervention. Maintain normal eating/nutritional behaviors.

INTERVENTIONS:
Behavioral: Virtual Reality Exergaming — The VR intervention will include home-based exercise using the Oculus Quest, a heart rate monitor (Polar OH1), BP cuff, and mobile application. The games will include rhythmic movements to music and sport/recreation activities that elicit high energy expenditure. Participants will be instructed to reach 150 minutes per week of moderate-exercise in week 1 and maintain this volume across the 12-week intervention. The intervention will include behavioral, physical education coaching through videoconference, which we refer to as Tele-PE. Tele-PE will aim to enhance adherence, provide basic exercise knowledge, and increase mastery playing the games. Calls will last 15 minutes, and be provided weekly in month 1, bi-weekly in month 2, and one call at the end of month 3.
  Arms: Immediate Start - Virtual Reality Exergaming

SUMMARY:
The primary purpose of this study is to examine the preliminary efficacy of 12-weeks of home-based exercise using consumer available virtual reality gaming technology, compared with a 12 week wait-list control group. The secondary purpose is to understand behavioral mechanisms that explain participation in exergaming through semi-structured interviews with participants from both groups at post-intervention or dropout.

DETAILED DESCRIPTION:
Youth with cerebral palsy (YwCP) do not have adequate exercise options that empower them to independently maintain their cardiometabolic health and, thus, live inactive, sedentary lifestyles that place them at substantially higher risk for cardiovascular disease, related conditions (e.g., hypercholesterolemia, diabetes, and hypertension), and mortality than the general population. No randomized controlled trial (RCT) has demonstrated clinically meaningful improvements in cardiometabolic health in people with cerebral palsy.

VR gaming delivered via telehealth may be an optimal method of promoting sustainable exercise behavior among large groups of youth. Home-based telehealth programs that incorporate 'virtual' behavioral coaching (tele-coaching) are a desirable approach for promoting non-supervised, exercise behavior among people with disabilities who do not have convenient access to community programs. The addition of behavioral coaching strategies such as goal-setting, confidence building, setting reasonable expectations, and understanding benefits, underpinned by theory such as the Social Cognitive Theory (Bandura, 2004), have been found to enhance the likelihood that people engage in and sustain a behavior.

Therefore, this study hypothesizes that 3-months of tele-monitored VR exergaming with behavioral coaching will result in strong adherence to moderate-intensity exercise and greater changes in key indicators of cardiometabolic health in YwCP, compared with a wait-list control group that maintains habitual activity (before receiving the intervention).

ELIGIBILITY:
Inclusion Criteria:

1. medical diagnosis of cerebral palsy
2. between the ages of 13-24 years to accommodate the World Health Organization definition of youth and the minimum age of 13 years specified by the Quest
3. physician clearance to participate
4. access to a Wi-Fi Internet connection in the home via mobile phone or tablet computer
5. a caregiver to support the child

Exclusion Criteria:

1. physically active (defined as >150 minutes per week of moderate-to-vigorous intensity exercise in a typical week)
2. cannot use their arms for exercise or a classification of GMFCS level V, which we have found to preclude the ability to use the Oculus Quest hand-held controllers
3. complete blindness or deafness.
4. contraindications to exercise based on the American College of Sports Medicine (ACSM) guidelines

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byron Lai, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be submitted into the NICHD Data and Specimen Hub (DASH). Intellectual property and data generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance under notice NOT-OD-03-032 (released February 26, 2003)
Supporting Information: Study Protocol
Time Frame: Beginning 3 months after publication and ending 5 years after publication.

REFERENCES:
- [Derived] Lai B, Davis D, Young R, Kimani-Swanson E, Wozow C, Wen H, Kim Y, Wilroy J, Rimmer J. The Effects of Virtual Reality Tele-exergaming on Cardiometabolic Indicators of Health Among Youth With Cerebral Palsy: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Aug 17;11(8):e40708. doi: 10.2196/40708. PMID 35976192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Started | 17 | 15
Completed | 13 | 15
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Children and youth with cerebral palsy
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (3.7) | 16.4 (3.8) | 16.7 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 15 | 10 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Gross Motor Function Classification System Level [Mean (Standard Deviation); unit: units on a scale] — A standardized 5-level classification system designed to describe the gross motor function of individuals with cerebral palsy:
  Scale Range:
  Level I: Walks without limitations.
  Level II: Walks with limitations.
  Level III: Walks using a hand-held mobility device.
  Level IV: Self-mobility with limitations; may use powered mobility.
  Level V: Transported in a manual wheelchair; limited in ability to maintain antigravity head and trunk postures.
  Higher values indicate poorer mobility.
  units on a scale | 2.18 (1.1) | 2.27 (1.1) | 2.22 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Changes in C-reactive Protein (hsCRP)
Description: hsCRP (mg/L) is a critical marker of inflammation that contributes to pro-inflammatory and pro-thrombotic elements of CVD risk. A single hsCRP measure is a strong predictor of myocardial infarction or coronary heart disease mortality, and several other diseases of the circulatory system in people without a history of such conditions.
Time Frame: Week 0
Population: Blood spot test
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/L | 2.32 (3.6) | 2.66 (3.5)

2. Primary Outcome: Changes in Hemoglobin A1C
Description: HbA1C (mmol/mol) measures mean hemoglobin glycation over the previous three months.
Time Frame: Week 0
Population: Blood spot test
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmol/mol | 4.51 (0.42) | 4.51 (0.55)

3. Primary Outcome: Changes in Fasting Insulin
Description: High fasting insulin indicates the presence of insulin resistance. Exercise interventions can expect a small beneficial change in fasting insulin levels after 1-month of training.
Time Frame: Week 0
Population: blood spot test
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
µIU/mL | 11.3 (5.7) | 11.6 (9.1)

4. Primary Outcome: Changes in Fasting Triglycerides
Description: A triglyceride level >150 mg/dL, is largely supported as an indicator of CVD risk. Exercise interventions can expect a small beneficial change in triglyceride levels following 1-month of training, even among people with normal triglyceride levels.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 102.1 (57.8) | 95.5 (41.9)

5. Primary Outcome: Changes in High-density Lipoprotein
Description: High-density lipoprotein (HDL; mg/dL) cholesterol is a predictor of future CVD among young and middle-aged people. Exercise interventions can expect a small effect after 1-month of training.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 46.6 (12.4) | 46.7 (10.8)

6. Primary Outcome: Changes in Low-density Lipoprotein
Description: Low-density lipoprotein (LDL; mg/dL) cholesterol is a predictor of future CVD among young and middle-aged people. Exercise interventions can expect a small effect after 1-month of training.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 112.8 (29.2) | 103.7 (28.8)

7. Primary Outcome: Changes in Total Cholesterol
Description: Total cholesterol (mg/dL) is a predictor of future CVD among young and middle-aged people. Exercise interventions can expect a small effect after 1-month of training.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 179.7 (34.7) | 169.5 (23.5)

8. Primary Outcome: Changes in Resting Systolic Blood Pressure
Description: Elevated blood pressure (mmHg) during childhood and adolescents is associated with intermediate markers and hard outcomes of CVD in adulthood. Moderate-intensity exercise is negatively associated with blood pressure. Small changes in blood pressure can occur from as early as 1-month of endurance training.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmHg | 106.1 (10.9) | 113.4 (14.8)

9. Primary Outcome: Changes in Resting Diastolic Blood Pressure
Description: as for outcome 8
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmHg | 71 (7.6) | 74.3 (8.5)

10. Primary Outcome: Changes in Body Weight
Description: Body weight measured in lbs using a off-the-shelf bathroom scale.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
lbs | 127.9 (42.3) | 128.5 (35.4)

11. Primary Outcome: Changes in Lung Capacity
Description: Lung capacity will be measured via peak expiratory flow rate (PEF; units: L/min) using a spirometer at the home.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
L/min | 323.71 (140) | 281.73 (87)

12. Primary Outcome: Changes in C-reactive Protein (hsCRP)
Description: as for outcome 1
Time Frame: Week 7
Population: Blood spot test
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/L | 2.91 (4) | 3.8 (3.8)

13. Primary Outcome: Changes in C-reactive Protein (hsCRP)
Description: as for outcome 1
Time Frame: Week 13
Population: Blood spot test
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/L | 9.1 (4.7) | 17.3 (18.7)

14. Primary Outcome: Changes in Hemoglobin A1C
Description: HbA1C (mmol/mol) measures mean hemoglobin glycation over the previous three months.
Time Frame: Week 7
Population: Blood spot test
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmol/mol | 4.68 (0.49) | 4.59 (0.48)

15. Primary Outcome: Changes in Hemoglobin A1C
Description: HbA1C (mmol/mol) measures mean hemoglobin glycation over the previous three months.
Time Frame: Week 13
Population: Blood spot test
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmol/mol | 4.7 (0.62) | 4.55 (0.47)

16. Primary Outcome: Changes in Fasting Insulin
Description: as for outcome 3
Time Frame: Week 7
Population: blood spot test
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
µIU/mL | 6.6 (2.4) | 15.6 (8.5)

17. Primary Outcome: Changes in Fasting Insulin
Description: as for outcome 3
Time Frame: Week 13
Population: blood spot test
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
µIU/mL | 9.1 (4.7) | 17.3 (18.7)

18. Primary Outcome: Changes in Fasting Triglycerides
Description: as for outcome 4
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 80 (28.4) | 100.7 (31.1)

19. Primary Outcome: Changes in Fasting Triglycerides
Description: as for outcome 4
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 90 (29.2) | 88.1 (33.9)

20. Primary Outcome: Changes in High-density Lipoprotein
Description: as for outcome 5
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 40.5 (9.3) | 49.6 (13)

21. Primary Outcome: Changes in High-density Lipoprotein
Description: as for outcome 5
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 43.1 (13) | 46.6 (12.9)

22. Primary Outcome: Changes in Total Cholesterol
Description: as for outcome 7
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 164.4 (30.7) | 168.4 (24.3)

23. Primary Outcome: Changes in Total Cholesterol
Description: as for outcome 7
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 176.8 (39.3) | 176.1 (35.7)

24. Primary Outcome: Changes in Low-density Lipoprotein
Description: as for outcome 6
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 107.3 (25) | 98.8 (24.6)

25. Primary Outcome: Changes in Low-density Lipoprotein
Description: as for outcome 6
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mg/dL | 117.2 (30.7) | 111.9 (32.2)

26. Primary Outcome: Changes in Resting Systolic Blood Pressure
Description: as for outcome 8
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmHg | 104.2 (10.6) | 111.3 (10)

27. Primary Outcome: Changes in Resting Systolic Blood Pressure
Description: as for outcome 8
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmHg | 103.2 (13.2) | 111.4 (14.8)

28. Primary Outcome: Changes in Resting Diastolic Blood Pressure
Description: as for outcome 8
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmHg | 71 (10.3) | 70.7 (7)

29. Primary Outcome: Changes in Resting Diastolic Blood Pressure
Description: as for outcome 8
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
mmHg | 70.3 (8.5) | 70.5 (7.9)

30. Primary Outcome: Changes in Body Weight
Description: Body weight measured in lbs using a off-the-shelf bathroom scale.
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
lbs | 127.7 (42) | 128.6 (36.7)

31. Primary Outcome: Changes in Body Weight
Description: Body weight measured in lbs using a off-the-shelf bathroom scale.
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
lbs | 128.1 (42.5) | 129 (38.4)

32. Primary Outcome: Changes in Lung Capacity
Description: Lung capacity will be measured via peak expiratory flow rate (PEF; units: L/min) using a spirometer at the home.
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
L/min | 316 (130) | 286 (103)

33. Primary Outcome: Changes in Lung Capacity
Description: Lung capacity will be measured via peak expiratory flow rate (PEF; units: L/min) using a spirometer at the home.
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 17 | 15
L/min | 359 (139) | 291 (109)

34. Secondary Outcome: Total Intervention Play Time
Description: Total minutes of playtime recorded by mobile app and uploaded to research staff by participants. Waitlist control data was not assessed for this outcome; data not collected.
Time Frame: Weeks 1-12
Population: These data were only analyzed from the immediate start group, not the control group.
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 13 | 0
minutes per week | 144 (73) |

35. Secondary Outcome: Adherence to the Exercise Intervention Prescription
Description: Percentage of moderate exercise minutes met (percent of prescription achieved), as indicated by participants in their exercise logs. The number of moderate minutes per week achieved divided by 150. Waitlist control data was not assessed for this outcome; data not collected.
Time Frame: Weeks 1-12
Population: Data were analyzed from only the immediate start group.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
Number analyzed (Participants) | 13 | 0
percentage | 64 (33) |

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: No participants had a serious adverse event. No participants were at risk for all-cause mortality, as the intensity of exercise was moderate and the participants were healthy (medically approved for exercise). The participant who had an adverse event was a unique case. He exercised in the standing position despite being prescribed to exercise in the seated position.
Arm/Group | Immediate Start - Virtual Reality Exergaming | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 1/17 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start - Virtual Reality Exergaming (N=17) | Wait-list Control (N=15)
Foot sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant played video game in the standing position. Due to high level of immersion, the participant kicked the wall and sprained their foot. The participant refrained from continuing the intervention for 3 weeks and withdrew.

LIMITATIONS AND CAVEATS:
The study sample was not statistically powered. Thus, findings should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT05336227/Prot_SAP_000.pdf